CLINICAL TRIAL: NCT04698551
Title: Comparison of Two NGS Phasing Techniques of Parental Haplotypes for NIPD of Triplet Expansion Diseases
Brief Title: NIPD on cffDNA for Triplet Repeat Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0441
Record Dates: First submitted 2020-09-01; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-09

CONDITIONS: Myotonic Dystrophy 1; Huntington Disease; Fragile X Syndrome
Keywords: Non Invasive Prenatal Diagnosis (NIPD); Circulating Fetal DNA (CFTC); triplet expansion diseases
MeSH Terms: conditions — Myotonic Dystrophy; Huntington Disease; Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 16 pregnant women and their spouses: 16 pregnant women and their spouses
  Interventions: Genetic: Non invasive prenatal diagnosis

INTERVENTIONS:
Genetic: Non invasive prenatal diagnosis — Search for the familial mutation involved in DPN requests from phasing of parental haplotypes by 3rd generation long-fragment DNA sequencing techniques coupled with targeted sequencing of free circulating DNA from maternal plasma.

SUMMARY:
The purprose of this study is to develop and validate an analytical NIPD test for triplet repeat disesases by NGS analysis from maternal blood, searching for the familial mutation in families at risk of having one of the following triplet repeat diseases: Huntington's disease, Myotonic dystrophy, Fragile X syndrome.. A comparison of two 3rd generation long fragment DNA sequencing techniques will be performed. These methods are based of the phasing techniques of parental haplotypes without the proband.

DETAILED DESCRIPTION:
Context:

The ability to sequence fetal cfDNA has led to exciting new developments for the non-invasive genetic diagnosis of monogenic diseases (DPNI_MGR). Various tests are proposed for diseases with predominantly de novo dominant, dominant paternal and some recessive paternal mutations. However, technical difficulties related to the determination of the maternal allelic balance remain, in particular during the phasing of parental haplotypes according to a trio strategy which requires the availability of parental genomic DNAs and at least one healthy or affected child. Moreover 2nd generation sequencers do not allow the haplotyping of alleles carrying dynamic mutations.

Objectives:

This project proposes the validation of a semi-universal DPNI_MGR test applicable to the majority of the genes and mutations involved in DPN requests from phasing of parental haplotypes by 3rd generation long-fragment DNA sequencing techniques coupled with targeted sequencing of free circulating DNA from maternal plasma. This test will be validated using triplet expansion diseases, which are the second indication of DPN at the national level.

Methodology :

Retrospective study of 16 couples at risk of transmitting a disease with triplet expansions (Myotonic dystrophy of Steinert, Huntington's disease, FRAXA, SCA1, 2, 3)

Phase 1 :

* Determination for 8 pairs of parental haplotypes according to the technique "Nanopore Cas9 Targeted-Sequencing" (nCATS) and validation of the analytical parameters and quality of this method (coverage rate of the regions of interest, error rate, identification of the morbid allele carrying the expansion ...),
* Comparison of the parental haplotypes obtained in "Nanopore" technique versus those obtained by the "Linked Reads 10xGenomics" technique in these same 8 pairs (the sequencing and phasing data by this 2nd approach are available from a previous study),
* Evaluation of the concordance of the fetal genotype results obtained during the standard examination (DPN by amniocentesis or choriocentesis) and those obtained with these new approaches of phasing in PNID.

Phase 2:

- Validation of the best performing workflow (efficiency / cost) of phase 1 over 8 additional pairs for a clinical transfer of the approach.

Expected results and prospects:

This study should make it possible to define the best performing test for the DPNI of triplet expansion diseases in accordance with the knowledge of the art and to validate the transfer conditions in clinical practice of the approach (equipment, reagents, cost analysis, analytical validation criteria ....).

The validated workflow should be as universal as possible to secondarily provide national level access to a wide range of rare diseases NIDP by future adjustments of the gene content of the free circulating DNA sequencing panels.

ELIGIBILITY:
Inclusion criteria:

* Couple at risk (based on family history or echographic findings) for one of the following diseases: Huntington's disease, Steinert's myotonic dystrophy, fragile X
* Written informed consent was obtained for DIACCIMEX study and mentionned "authorization for use for further studies on familial pathology. Indeed, the DNA can be used anonymized for the development of new analyzes of non-invasive prenatal diagnosis".
* Prenatal diagnosis has been done for the pregnancy during which maternal blood has been collected
* Couple molecular diagnosis results for one of the following diseases (Huntington's disease, Steinert's myotonic dystrophy, fragile X and spinocerebellar ataxias 1, 2 or 3 ) MUST BE AVAILABLE.

Exclusion criteria:

* Couple Genomic DNA are unavailable
* Subjects at risk of transmitting the family disease, but not wishing to know their molecular status
* Individuals under guardianship by court order

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective study of 16 couples at risk of transmitting a disease with triplet expansions (Myotonic dystrophy of Steinert, Huntington's disease, FRAXA) Couples undergoing prenatal diagnosis for a monogenic disease caused by dynamic mutation
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Concordance rate between cell free foetal DNA based genetic | 36 months
  t is a qualitative analysis : for each sample of each pregnant women, the presence of absence of a mutation (or morbid haplotype) responsible for a triplet expansion will be determined from maternal blood (Non invasive Pregnancy Diagnosis). the result could be : health fetus, affected fetus or non conclusive result (i.e. the analysis didn't allow to conclude if the fetus would be affected or not) Then, determination of the concordance rate between cell-based genetic non invasive prenatal test and gold standard prenatal test (choriocentesis or amniocentesis). Analysis of the concordance of the prenatal results obtained by our new NIPD (Non-Invasive Prenatal Diagnosis) approach and those blindly obtained during the gold-standard prenatal genetic test will be carried out for each pregnant woman participating in the study

SECONDARY OUTCOMES:
Qualitative process to define the differents steps to analysis of the cell free foetal DNA | 36 months
  Qualitative choice : define the most efficiency workflow in term of ratio cost/efficacity between the two kits of long fragment sequencing (simplicity, rapidity, accuracy and cost of the products )

CONTACTS AND LOCATIONS:
Overall Officials: Marie Claire VINCENT, PhD-PharmaD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Liautard-Haag C, Durif G, VanGoethem C, Baux D, Louis A, Cayrefourcq L, Lamairia M, Willems M, Zordan C, Dorian V, Rooryck C, Goizet C, Chaussenot A, Monteil L, Calvas P, Miry C, Favre R, Le Boette E, Fradin M, Roux AF, Cossee M, Koenig M, Alix-Panabiere C, Guissart C, Vincent MC. Noninvasive prenatal diagnosis of genetic diseases induced by triplet repeat expansion by linked read haplotyping and Bayesian approach. Sci Rep. 2022 Jul 6;12(1):11423. doi: 10.1038/s41598-022-15307-2. PMID 35794169